CLINICAL TRIAL: NCT00915941
Title: Exploratory Study of Potential Pulmonary Aspiration Markers From Bronchoalveolar Lavage Fluid"
Brief Title: Exploratory Study of Potential Pulmonary Aspiration Markers From Bronchoalveolar Lavage Fluid
Acronym: Pepsin
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. Augustine Lee, Mayo Clinic Florida
Other Study IDs: 07-000550
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BALF specimens will be collected by the MCF Biospecimen Facility at the time of the bronchoscopy. A minimum of 5 mL will be collected. Specimen processing will include centrifugation to separate the cell pellet from the supernatant. The supernatant will be stored in 2 mL cryovials, and stored at -70°C until time of testing for the pepsin-ELISA. Storage will allow retesting at another date if the assay is modified or if another substance of interest arises in the course of the study that requires re-testing of the specimens. The clinical sample will also be tested through the Mayo Clinic medical laboratory for bilirubin, pepsinogen, amylase, and lipase.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn if chemicals from the mouth or stomach can be found in the lungs. This may suggest a process called aspiration. This study may help us understand if aspiration plays a role in different lung diseases.

DETAILED DESCRIPTION:
This study is a single center, prospective, observational study of determining pepsin levels in BALF samples obtained from consecutive bronchoscopies at the Mayo Clinic Jacksonville. It is inherently an exploratory pilot study to confirm whether pepsin in BAL can act as a marker of gastric to pulmonary aspiration and whether specific association to pulmonary pathologies can be identified.

As an overview, all patients who are undergoing a bronchoscopy for clinical indications will be screened for potential participation in the study by obtaining BALF samples during the procedure for laboratory analyses. The BALF will then be tested for pepsin at the Thoracic Diseases Research Unit (Mayo Clinic Rochester) using a commercially available ELISA kit, and the ancillary markers will be analyzed per the clinical laboratory. Internal controls will be defined as normals when subjects have no lung dysfunction, no respiratory symptoms, and no lung parenchymal infiltrates on chest radiographs.

The primary aims of this project parallels the short-term hypotheses stated above:

1. Confirm pepsin can be detected and quantitated in BALF obtained during a routine bronchoscopy.
2. Identify specific pulmonary pathologies that are more often associated with increased pepsin BAL levels.
3. Identify a normal range of pepsin in BALF in control normals.
4. Identify any correlation of pepsin BAL levels with reflux, swallow, or respiratory symptoms (standardized questionnaires).
5. Identify any correlation between pepsin BAL levels and lung function test or radiographic abnormalities.

Secondary aims of the study will include exploratory analyses of lesser defined potential aspiration markers including bilirubin, lipase, amylase, and pepsinogen. Analyses of these markers will parallel the analyses performed for pepsin.

The focus of the study is to:

* definitively identify whether pulmonary aspiration is occurring;
* quantitate the burden of aspiration that is occurring (i.e., dose);
* localize from where aspiration is occurring (e.g., gastric, duodenal, biliary, oropharyngeal, nasal);
* identify what is specifically being aspirated (e.g., acid, exogenous oils, bacteria, gastric contents, bile, gastric enzymes, pancreatic enzymes).

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing bronchoscopy for clinical reasons
2. 21 years of age or older
3. Ordering clinician and bronchoscopist is consenting

Exclusion Criteria:

1. Emergent bronchoscopies
2. Bronchoscopies performed in the operating room
3. Pre-procedural oxygen requirement > 2 LPM for those who do not have a bronchoalveolar lavage ordered by the clinician as part of the bronchoscopy
4. Pre-procedural bronchospasm for those who do not have a bronchoalveolar lavage ordered by the clinician as part of the bronchoscopy
5. BAL is not requested for clinical reasons in a hospitalized or a mechanically ventilated patient
6. The study coordinator, investigator, clinician, or the bronchoscopist may at any time withdraw the patient with regards to any concerns on patient safety or if there is concerns on the patient's or patient's surrogate's ability to give an informed consent
7. The clinician or the bronchoscopist may at any time withdraw the patient if by participating in the study, the bronchoalveolar fluid obtained is felt to be inadequate for clinical testing

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be recruited from the Mayo Clinic Jacksonville site. As defined in the inclusion criteria, patients will only be identified once they are scheduled for a bronchoscopy for clinical indications. Only adult patients will be considered, and there will be no regard to gender or ethnicity in the screening or selection. The BAL procedure may or may not be requested by the referring clinician as part of the patient's bronchoscopy. In those subjects where the BAL is not requested for clinical indications, that means the BAL will be an additional procedure to be added to the patient's bronchoscopy for research purposes. Both patients in the inpatient and outpatient settings will be recruited, but emergent or operating room based bronchoscopies will be excluded. The specific inclusion and exclusion criteria are listed below.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States